CLINICAL TRIAL: NCT04738266
Title: A National Survey of Prevalence and Accuracy of Echocardiographic Red Flags of Amyloid Cardiomyopathy in Consecutive Patients Undergoing Routine Echocardiography.
Brief Title: Unmasking the Prevalence of AC in an Unselected Echocardiographic Population
Acronym: AC-TIVE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Trieste (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Marco Merlo, MD, Associate Professor, University of Trieste
Other Study IDs: 199_2019
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Amyloid Cardiomyopathy
Keywords: Amyloid Cardiomyopathy; Echocardiography; Red flags; Epidemiology; Bone tracer cardiac scintigraphy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Amyloid Cardiomyopathy — Echocardiographic red flags of Amyloid Cardiomyopathy to guide the suspicion of disease and to proceed with second level diagnostic work up including cardiac scintigraphy with bone tracers and search of monoclonal component in serum and urine

SUMMARY:
This study will investigate the prevalence of echocardiographic red-flags of amyloid cardiomyopathy (AC) in patients undergoing clinically-indicated echocardiography (observational phase) and the prevalence of AC among AC-suggestive echocardiograms (interventional phase).

DETAILED DESCRIPTION:
Prospective multicenter Italian survey consisting of two phases: observational (echocardiographic screening for amyloid cardiomyopathy among patients ≥ 55 years undergoing clinically-indicated echocardiography) and interventional (specific clinical and instrumental work-up to detect the prevalence of amyloid cardiomyopathy among amyloid cardiomyopathy-suggestive echocardiograms).

ELIGIBILITY:
Inclusion Criteria:

All the following:

* Interventricular septum thickness ≥ 13 mm in men and ≥ 12 mm in women;
* Left ventricular ejection fraction ≥ 50%;
* Indexed end-diastolic left ventricular volume ≤ 85 mL/m2.

AND

At least one of the following criteria:

* "Granular sparkling" appearance of the myocardium defined granular texture with uniform increased brightness of echo-reflections;
* Pericardial effusion regardless of severity;
* Increased interatrial septum thickness (> 5 mm);
* Restrictive filling pattern (Dec. Time E wave <120 ms or Dec. Time E wave ≤150 ms e E/A ratio ≥2) or increased ventricular filling pressures (E/E'15);
* Speckle tracking derived global longitudinal strain with apical sparing pattern;
* Increased thickness (> 5 mm) of mitral and tricuspid valve leaflets.

Exclusion Criteria:

* Patients aged < 55 years or > 100 years
* Echocardiography performed due to known or suspected amyloid cardiomyopathy;
* Echocardiography performed due to known hypertrophic cardiomyopathy or phenocopies;
* Refuse to sign the informed consent to the study

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive inpatients and outpatients subjects aged ≥55 years undergoing routine, clinically-indicated echocardiography at the laboratories of participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
The prevalence of Amyloid Cardiomyopathy | 3 months
  The prevalence of Amyloid Cardiomyopathy in unselected echocardiographic population of patients aged > 55 years
The prevalence of echocardiographic red flags of Amyloid Cardiomyopathy | 6 months
  The prevalence of echocardiographic red flags of Amyloid Cardiomyopathy in unselected echocardiographic population of patients aged > 55 years
The diagnostic accuracy of echocardiographic red flags of Amyloid Cardiomyopathy | 6 months
  At the end of phase 2 of this study, patients with Amyloid Cardiomyopathy will be diagnosed, thus allowing to measure the diagnostic accuracy of the following echocardiographic red flags of Amyloid Cardiomyopathy:
  * Restrictive filling pattern (E wave deceleration time <120 ms or ≤150 ms in presence of E/A ≥2) and/or E/E'≥15;
  * "Granular sparkling" appearance of the myocardium;
  * Pericardial effusion of any entity;
  * Interatrial septum thickness >0.5 cm measured in subcostal or four-chamber view;
  * Thickening of the atrio-ventricular (AV) valves (leaflets thickness >0.5 cm);
  * Left ventricular "apical sparing" pattern at speckle-tracking echocardiography.

SECONDARY OUTCOMES:
Multiparametric echocardiographic score | 6 months
  Multiparametric echocardiographic score to predict the presence of Amyloid Cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Sinagra, MD, Full Professor, Study Chair — Azienda Sanitaria Universitaria Giuliano-Isontina (ASUGI) and University of Trieste; Claudio Rapezzi, MD, Full Professor, Study Chair — Cardiology Unit, Azienda Ospedaliero Universitaria di Ferrara - Ferrara
Locations (16):
- Italy (16):
  - Emergency Department and Amyloid Research and Treatment Center, IRCCS Policlinico San Matteo Foundation, Department of Internal Medicine, University of Pavia, Pavia, Milano
  - Cardiology Unit, Department of Emergency and Organ Transplantation, University of Bari Aldo Moro, Bari
  - Cardiovascular Department, Policlinico Sant'Orsola, Bologna
  - Cardiology, Department of Medical and Surgical Specialities, Radiological Sciences and Public Health - University of Brescia, Brescia
  - Cardiology Unit, Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - Cardiomyopathy Unit, Careggi University Hospital, Florence
  - Cardiovascular Unit, Department of Internal Medicine, University of Genova, Genova
  - Department of Cardiology, University of Messina, Messina
  - Department of medicine and surgery, University Milano-Bicocca, Milan
  - Department of Cardiovascular, Neural and Metabolic Sciences - Istituto Auxologico Italiano, Milan
  - Department of Translational Medical Sciences, Inherited and Rare Heart Disease, Vanvitelli Cardiology, University of Campania Luigi Vanvitelli, Napoli
  - Istituto di Scienze della Vita, Scuola Superiore Sant'Anna, Pisa
  - Department of Clinical and Molecular Medicine, Faculty of Medicine and Psychology, Sapienza University, Roma
  - Division of Cardiology, University of Siena, Siena
  - University Cardiology A.O.U., Città della Salute e della Scienza di Torino, Torino
  - Centre for Diagnosis and Treatment of Cardiomyopathies, Cardiovascular Department, Azienda Sanitaria Universitaria Giuliano-Isontina (ASUGI), Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maurer MS, Bokhari S, Damy T, Dorbala S, Drachman BM, Fontana M, Grogan M, Kristen AV, Lousada I, Nativi-Nicolau J, Cristina Quarta C, Rapezzi C, Ruberg FL, Witteles R, Merlini G. Expert Consensus Recommendations for the Suspicion and Diagnosis of Transthyretin Cardiac Amyloidosis. Circ Heart Fail. 2019 Sep;12(9):e006075. doi: 10.1161/CIRCHEARTFAILURE.119.006075. Epub 2019 Sep 4. PMID 31480867
- [Background] Boldrini M, Cappelli F, Chacko L, Restrepo-Cordoba MA, Lopez-Sainz A, Giannoni A, Aimo A, Baggiano A, Martinez-Naharro A, Whelan C, Quarta C, Passino C, Castiglione V, Chubuchnyi V, Spini V, Taddei C, Vergaro G, Petrie A, Ruiz-Guerrero L, Monivas V, Mingo-Santos S, Mirelis JG, Dominguez F, Gonzalez-Lopez E, Perlini S, Pontone G, Gillmore J, Hawkins PN, Garcia-Pavia P, Emdin M, Fontana M. Multiparametric Echocardiography Scores for the Diagnosis of Cardiac Amyloidosis. JACC Cardiovasc Imaging. 2020 Apr;13(4):909-920. doi: 10.1016/j.jcmg.2019.10.011. Epub 2019 Dec 18. PMID 31864973
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678
- [Background] Maurer MS, Elliott P, Comenzo R, Semigran M, Rapezzi C. Addressing Common Questions Encountered in the Diagnosis and Management of Cardiac Amyloidosis. Circulation. 2017 Apr 4;135(14):1357-1377. doi: 10.1161/CIRCULATIONAHA.116.024438. PMID 28373528
- [Background] Porcari A, Merlo M, Rapezzi C, Sinagra G. Transthyretin amyloid cardiomyopathy: An uncharted territory awaiting discovery. Eur J Intern Med. 2020 Dec;82:7-15. doi: 10.1016/j.ejim.2020.09.025. Epub 2020 Oct 5. PMID 33032855
- [Background] Maurer MS, Hanna M, Grogan M, Dispenzieri A, Witteles R, Drachman B, Judge DP, Lenihan DJ, Gottlieb SS, Shah SJ, Steidley DE, Ventura H, Murali S, Silver MA, Jacoby D, Fedson S, Hummel SL, Kristen AV, Damy T, Plante-Bordeneuve V, Coelho T, Mundayat R, Suhr OB, Waddington Cruz M, Rapezzi C; THAOS Investigators. Genotype and Phenotype of Transthyretin Cardiac Amyloidosis: THAOS (Transthyretin Amyloid Outcome Survey). J Am Coll Cardiol. 2016 Jul 12;68(2):161-72. doi: 10.1016/j.jacc.2016.03.596. PMID 27386769
- [Derived] Merlo M, Pagura L, Porcari A, Cameli M, Vergaro G, Musumeci B, Biagini E, Canepa M, Crotti L, Imazio M, Forleo C, Cappelli F, Perfetto F, Favale S, Di Bella G, Dore F, Girardi F, Tomasoni D, Pavasini R, Rella V, Palmiero G, Caiazza M, Carella MC, Igoren Guaricci A, Branzi G, Caponetti AG, Saturi G, La Malfa G, Merlo AC, Andreis A, Bruno F, Longo F, Rossi M, Varra GG, Saro R, Di Ienno L, De Carli G, Giacomin E, Arzilli C, Limongelli G, Autore C, Olivotto I, Badano L, Parati G, Perlini S, Metra M, Emdin M, Rapezzi C, Sinagra G. Unmasking the prevalence of amyloid cardiomyopathy in the real world: results from Phase 2 of the AC-TIVE study, an Italian nationwide survey. Eur J Heart Fail. 2022 Aug;24(8):1377-1386. doi: 10.1002/ejhf.2504. Epub 2022 May 10. PMID 35417089